CLINICAL TRIAL: NCT03775317
Title: Comparison of Video-assisted Laryngoscopy and Direct Laryngoscopy for Routine Nasotracheal Intubation in Oral and Maxillofacial Surgery Patients: a Randomized Controlled Trial.
Brief Title: Video Laryngoscopy Versus Direct Laryngoscopy for Nasotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Brett King, Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10272
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Intubation, Intratracheal
Keywords: Video laryngoscopy; Nasal intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Laryngoscopy (Experimental)
  Interventions: Procedure: Video Laryngoscopy
- Direct Laryngoscopy (Active Comparator)
  Interventions: Procedure: Direct Laryngoscopy

INTERVENTIONS:
Procedure: Video Laryngoscopy — The direct, or conventional, laryngoscopy group will undergo the planned nasotracheal intubation utilizing a Macintosh or Miller laryngoscope for direct visualization of the larynx.
  Arms: Video Laryngoscopy
Procedure: Direct Laryngoscopy — The video-assisted laryngoscopy group will undergo the planned nasotracheal intubation utilizing a Storz C-MAC S Video Laryngoscope to allow for indirect visualization of the larynx.
  Arms: Direct Laryngoscopy

SUMMARY:
Nasotracheal intubation is a common method for securing an advanced airway during surgery for procedures that involve manipulation of the oral cavity, the dentition, or the facial bones. The placement of a nasotracheal tube is often more challenging, especially for learning providers, even for patients with normal airway anatomy. Video laryngoscopy is an adjunctive technique in anesthesia that utilizes a camera at the tip of the laryngoscope blade and provides an indirect view of the glottis during intubation through display on a monitor. The use of video laryngoscopes has been shown to reduce time to intubation, result in perception of easier intubation by the anesthesia team, and reduce the use of adjunctive maneuvers during intubation. There is little evidence, however, to show these benefits for routine nasotracheal intubation. The purpose of the study is to compare the ease of video-assisted laryngoscopy and direct laryngoscopy in routine nasotracheal intubation for Maxillofacial procedures. The investigators hypothesize that the use of video-assisted laryngoscopy for routine nasotracheal intubation will result in quicker time to intubation, less adjunctive maneuvers and anesthesia perception of easier intubation when compared to direct nasotrahceal intubation. The investigators aim to compare the time to intubation, number of adjunctive maneuvers and the perception of intubation difficulty in routine nasotracheal intubation for Maxillofacial procedures for video-assisted laryngoscopy and direct laryngoscopy.

DETAILED DESCRIPTION:
Comparison of video-assisted laryngoscopy and direct laryngoscopy for routine nasotracheal intubation in oral and maxillofacial surgery patients: a randomized controlled trial.

INTRODUCTION Nasotracheal intubation is a common method for securing an advanced airway during surgery for procedures that involve manipulation of the oral cavity, the dentition, or the facial bones. The placement of a nasotracheal tube is often more challenging, especially for learning providers, even for patients with normal airway anatomy. Video laryngoscopy is an adjunctive technique in anesthesia that utilizes a camera at the tip of the laryngoscope blade and provides an indirect view of the glottis during intubation through display on a monitor. The use of video laryngoscopes has been shown to reduce time to intubation, result in perception of easier intubation by the anesthesia team, and reduce the use of adjunctive maneuvers during intubation. There is little evidence, however, to show these benefits for routine nasotracheal intubation. The purpose of the study is to compare the ease of video-assisted laryngoscopy and direct laryngoscopy in routine nasotracheal intubation for Maxillofacial procedures. The investigators hypothesize that the use of video-assisted laryngoscopy for routine nasotracheal intubation will increase the rate of success on first intubation attempt, result in quicker time to intubation, less adjunctive maneuvers and anesthesia perception of easier intubation when compared to direct nasotrahceal intubation. The investigators aim to compare the rate of first attempt intubation success, time to intubation, number of adjunctive maneuvers and the perception of intubation difficulty in routine nasotracheal intubation for Maxillofacial procedures for video-assisted laryngoscopy and direct laryngoscopy.

METHODS Study Sample After obtaining institutional review board approval (IRB #10272), the authors will design a randomized clinical trial. The eligible study population will include all patients who presented to University Medical Center in New Orleans, LA for oral and maxillofacial surgery to be performed under general anesthesia and planned for a nasotracheal intubation. The inclusion criteria for the study will be as follows: planned for a general anesthetic with nasotracheal intubation, ASA I and II and at least 18 years of age. Prisoners and patients with anticipated difficult airways will be excluded from this study.

Study Design This will be a single center, parallel group, unblinded randomized controlled trial with an allocation ratio of 1:1. Because the investigators hypothesized that video-assisted laryngoscopy would increase the rate of success of intubation on the first attempt and previous data shows this trend in a similar patient population (Tabrizi et al 2018), this trial will be designed to assess for superiority of the video-assisted laryngoscopy. One of the investigators will explain the risks and benefits of participation in the study in detail to each patient and patients will be enrolled in the study after signing informed consent. A co-investigator, not involved with enrollment or the anesthetic, will use a computerized research randomization software (www.randomizer.org) to perform block randomization with randomly varying block sizes of 2, 4 and 6. Then, he will place a paper with the group allocation written on it into sequentially numbered envelopes in the order determined by the randomization software. The group allocation will be concealed by using opaque envelopes that will be sealed after the paper with the group assignment is placed in the envelope. When a patient is enrolled in the study, the next envelope in the sequence will be labeled with the patient's study ID and opened by the principal investigator, who ensured the anesthetic team then performed the technique for intubation assigned to the patient. The direct, or conventional, laryngoscopy group will undergo the planned nasotracheal intubation utilizing a Macintosh or Miller laryngoscope for direct visualization of the larynx. The video-assisted laryngoscopy group will undergo the planned nasotracheal intubation utilizing a Storz C-MAC S Video Laryngoscope to allow for indirect visualization of the larynx.

Variables The primary outcome variable will be the success of first attempt intubation. Success of intubation will be defined as confirmed placement of the endotracheal tube by bilateral breath sounds, end-tidal CO2 waveform and lack of cuff leak. The secondary outcome variables will be the amount of time required to secure the nasotracheal tube, the use of Macgill forceps, the success at first attempt, the number of attempts, the number of endotracheal tube exchanges after placement and the number of torn endotracheal tube cuffs. Time for intubation will be recorded for each case by an independent observer using a stopwatch which will start upon removal of the bag mask and will end after the anesthesiologist confirmed bilateral breath sounds, an end-tidal CO2 waveform and lack of cuff leak. Use of Macgill forceps will be recorded by an independent observer upon their use during intubation. An attempt at intubation will be considered failed when the laryngoscope is removed from the mouth prior to insertion of the endotracheal tube and bask mask ventilation is restarted. Tube exchanges will likewise be recorded if they occur.

The predictor variable will be the laryngoscopy technique employed: video-assisted laryngoscopy (the experimental group) or direct Macintosh or Miller laryngoscopy (the control group). Other variables that will be recorded are age, gender, ASA score and procedure performed.

Sample Size Calculation The sample size for the study was calculated based on a difference of 10% in first attempt success rate between groups. The investigators regarded this amount of time as the smallest meaningful difference. Previously published reports was used to base the sample size calculation, using a success rate of 82% and 60% for first attempt at video laryngoscopy and direct laryngoscopy, respectively. An estimated sample size of 48 patients (24 in each arm) will be needed to detect a difference of 10% in first attempt success rate between the groups with an 80% power and alpha level of 0.05. [A previously published study (Rabrizi et al 2018) assessed first attempt success rate in patients with bilateral mandibular fractures in Glidescope video laryngoscopy versus Macintosh laryngoscopy. They found a first attempt success rate of 82% using a video laryngoscopy versus 60% using direct laryngoscopy.] Data Collection and Analysis To organize data collection, a Microsoft Excel spreadsheet will be created and used to record information, which will be kept on a secured LSU drive which only the investigators have access to. Data will be compiled and imported into JMP Statistical Discovery for analysis (JMP, Version 12.1. SAS Institute Inc., Cary, NC, 1989-2015). The relationship of the primary outcome variable to the primary predictor will be analyzed using Chi squared tests. The relationship of the secondary outcome variables to the primary predictor will be analyzed using Chi squared tests and t tests, as appropriate for the data type. Study variables will be examined for their relationship to the primary predictor and primary outcome using t test, Chi squared test and ANOVA as appropriate for the type of variable. A p-value of less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* oral and maxillofacial surgery to be performed under general anesthesia
* planned for a general anesthetic with nasotracheal intubation,
* ASA I and II
* at least 18 years of age

Exclusion Criteria:

* prisoners
* anticipated difficult airways

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
success of first attempt intubation | 1 day
  defined as confirmed placement of the endotracheal tube by bilateral breath sounds, end-tidal CO2 waveform and lack of cuff leak

SECONDARY OUTCOMES:
amount of time required to secure the nasotracheal tube | 1 day
  amount of time required to secure the nasotracheal tube
the use of Macgill forceps | 1 day
  the use of Macgill forceps
success at first attempt | 1 day
  success at first attempt
number of attempts | 1 day
  number of attempts
number of endotracheal tube exchanges after placement | 1 day
  number of endotracheal tube exchanges after placement
number of torn endotracheal tube cuffs | 1 day
  number of torn endotracheal tube cuffs
Cormack-Lehane score | 1 day
  Cormack-Lehane score

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No